CLINICAL TRIAL: NCT04689412
Title: Intermittent Treatment With Nasal Resveratrol and Reduction of Wheezing Episodes in Non Atopic Preschool Children
Brief Title: Nasal Resveratrol and Wheezing Episodes in Preschool Children
Acronym: RSVchild
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Giuseppe Di Cara, PhD, MD, Prof. Giuseppe Di Cara, University Of Perugia
Other Study IDs: RSV01Ped
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Wheezing; Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Sounds; Respiratory Tract Infections | interventions — Resveratrol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children spontaneously treated with nasal resveratrol at the beginning of each upper airways infection
  Interventions: Drug: Resveratrol
- Controls: Children spontaneously treated with nasal lavage at the beginning of each upper airways infection

INTERVENTIONS:
Drug: Resveratrol — Nasal administration of resveratrol
  Groups: Cases

SUMMARY:
As most of the upper airways infections (UAI) leading to wheezing are secondary to viral triggers, the possible antinflammatory and antiviral role of resveratrol has been suggested in several studies, both in vitro and in vivo. However, its efficacy has been studied only when evaluating upper respiratory symptoms.

With the aim to define new approaches in patients with recurrent wheezing triggered by UAI we have performed a prospective observational study to evaluate the efficacy of a short-course of intranasal resveratrol, administered for 7 days at the beginning of UAI, when compared to standard nasal lavage with 0.9% saline solution, in terms of reduction in wheezing episodes.

DETAILED DESCRIPTION:
Patients Patients were selected from those referring to our centre for recurrent wheezing in the previous year.

The inclusion criteria were:

* Presence of at least 8 episodes of wheezing in the previous October-March period
* Negative skin prick test (SPT) for the most common allergens.
* Age less than 6 years

The exclusion criteria were:

* Sensitization to food allergens
* Sensitization to perennial allergens or to tree pollen allergens.
* Presence of atopic dermatitis

Patients were enrolled during visit 1, from April to August 2018, and were instructed to record symptoms of upper and lower airways during the wash-out period of September. During visit 2 at the end of September patients were randomized into 2 groups:

* group 1: patients treated with 0.9% saline solution daily nasal lavage
* group 2: patients treated with 0.9% saline solution daily nasal lavage and a 7-days therapy with nasal resveratrol, from the beginning of upper airways symptoms.

All patients were followed from September 2018 to the end of March 2019, with visit 3 and 4 after two (end of November) and four months (end of January). Follow-up ended with visit 5 at the end of March. All patients were instructed to register in specifically designated charts the number of days with symptoms of upper airways inflammation and the recurrence of wheezing. As predictive index of disease severity, parents were instructed to register both days with oral corticosteroids administration (OCA) and with hospitalization need, as ER occurrence or admission to paediatric wards. All patient were instructed to treat each wheezing episode with inhaled salbutamol and, if wheezing persisted, with oral prednisolone once a day, according to guidelines (Gina 2015).

Skin prick tests The sensitization status of each patient was assessed by performing skin prick tests (SPTs) with a standard panel of environmental (Stallergenes, Antony, France) and food allergens (Lofarma, Milan, Italy). Positivity of SPT was established according to the guidelines of the European Academy of Allergology and Clinical Immunology. The standard panel of allergens included Phleum pratense, Parietaria judaica, Juniperus ashei, Olea europaea, Dermatophagoides pteronyssinus, Alternaria tenuis, cat and dog epithelium; milk, egg, peanut, tree nuts, fish, shellfish, soy, and wheat plus a positive (histamine 10 mg/mL) and a negative (normal saline) control. Wheals were contoured with a soft pen and transferred onto cellotape. A skin reaction of 5 mm was considered the threshold for positivity.

Clinical symptoms, rescue medication and severity evaluation During the evaluation period, patients filled in daily diary cards to record days with symptoms involving the upper (sneezing, rhinorrhoea, itching and nasal blockage) and lower airways (cough, dyspnoea and wheezing), the use of oral corticosteroids (OCS) and the days of hospitalization when occurred.

ELIGIBILITY:
The inclusion criteria were:

* Presence of at least 8 episodes of wheezing in the previous October-March period
* Negative skin prick test (SPT) for the most common allergens.
* Age less than 6 years

The exclusion criteria were:

* Sensitization to food allergens
* Sensitization to perennial allergens or to tree pollen allergens.
* Presence of atopic dermatitis

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients were selected from those referring to our centre for recurrent wheezing in the previous year.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Wheezing days | october 2017 - march 2018
  number of wheezing days during the follow-up period

SECONDARY OUTCOMES:
Severity index | october 2017 - march 2018
  oral corticosteroid administration
Severity index | october 2017 - march 2018
  access to ER or admission to pediatric ward

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No